CLINICAL TRIAL: NCT04894045
Title: Perioperative Personalized Blood Pressure Management in Patients Having Major Surgery: a Bicentric Prospective Randomized Controlled Interventional Pilot Trial (IMPROVE-pilot)
Brief Title: Perioperative Personalized Blood Pressure Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-10462-BO-bet
Record Dates: First submitted 2021-04-24; First posted 2021-05-20 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Blood Pressure; Intraoperative Hypotension; Postoperative Complications
Keywords: Blood Pressure; Intraoperative Hypotension; Cardiovascular Dynamics
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In control group patients, the treating anesthesiologists are blinded to the data of preoperative automated blood pressure monitoring. Participants and outcomes assessors are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized management group (Other): Intraoperative MAP will be maintained at least at the mean nighttime MAP (assessed using preoperative automated blood pressure monitoring). If the mean nighttime MAP is below 65 mmHg, intraoperative MAP will be maintained at least at 65 mmHg.
  Interventions: Other: Personalized management
- Control group (No Intervention): Routine intraoperative blood pressure management with a lower intervention threshold of 65 mmHg. In contrast to the patients in the personalized management group, the individual mean nighttime MAP assessed using preoperative automated blood pressure monitoring is not taken into account and the treating anesthesiologists are blinded to the data of preoperative automated blood pressure monitoring.

INTERVENTIONS:
Other: Personalized management — Intraoperative MAP will be maintained at least at the mean nighttime MAP (assessed using preoperative automated blood pressure monitoring). If the mean nighttime MAP is below 65 mmHg, intraoperative MAP will be maintained at least at 65 mmHg.
  Arms: Personalized management group

SUMMARY:
The investigators propose a pilot trial to (1) proof the concept that defining the intraoperative mean arterial pressure (MAP) intervention threshold based on the mean nighttime MAP (assessed using preoperative automated blood pressure monitoring) results in clinically relevant (mean nighttime MAP ± 10 mmHg) different target values compared with using an absolute population-derived MAP intervention threshold of 65 mmHg (primary endpoint); (2) investigate if a personalized perioperative blood pressure management is feasibly in multi-center studies, especially if the target values can be sufficiently achieved (secondary endpoint); (3) study the impact of personalized perioperative blood pressure management on the incidence of myocardial injury after non-cardiac surgery (MINS) (exploratory endpoint); (4) study the impact of personalized perioperative blood pressure management on the incidence of acute kidney injury within the first three postoperative days according to the KDIGO (Kidney Disease: Improving Global Outcomes) definition without oliguric criteria (exploratory endpoint).

DETAILED DESCRIPTION:
not provided

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45
* American Society of Anesthesiologists physical status class (ASA) II-IV
* scheduled for elective major surgery under general anesthesia
* surgery expected to last ≥ 120 minutes

Exclusion Criteria:

* emergency surgery
* patients having liver or kidney transplantation
* laparoscopic surgery
* pregnancy
* status of post transplantation of kidney, liver, heart, or lung
* sepsis (according to current Sepsis-3 definition)
* impossibility of preoperative automated blood pressure monitoring
* MAP differences between the right and the left arm of more than 20 mmHg surgery that requires controlled hypotension

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
Individualized MAP target value | 1 day before surgery
  Difference between intraoperative target MAP (defined as the mean nighttime MAP assessed using preoperative automated blood pressure monitoring) and 65 mmHg; we consider a difference > ± 10 mmHg as clinically meaningful.

SECONDARY OUTCOMES:
Proportion of patients with calculated MAP target | day of surgery
  - proportion of patients in whom preoperative automated blood pressure monitoring + calculation of target MAP is possible
Duration and severity of MAP below MAP target | day of surgery
  - time weighted average MAP below individual MAP target

OTHER OUTCOMES:
Incidence of myocardial injury after non-cardiac surgery | baseline, postoperative days 1, 2 and 3
  Incidence of myocardial injury after non-cardiac surgery assessed through measurement of baseline high-sensitivity troponin T (before surgery) and high-sensitivity troponin T on postoperative days 1,2, and 3.
Incidence of acute kidney injury | baseline, postoperative day 1, 2 and 3
  Incidence of acute kidney injury within the first three postoperative days according to the KDIGO definition without oliguric criteria assessed through measurement of baseline creatinine (before surgery) and creatinine after surgery on postoperative days 1, 2, and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Saugel, Prof. Dr., Principal Investigator — Department of Anesthesiology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany; Karim Kouz, Dr., Principal Investigator — Department of Anesthesiology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany
Locations (2):
- Germany (2):
  - University Hospital RWTH Aachen, Aachen
  - Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Sessler DI, Bloomstone JA, Aronson S, Berry C, Gan TJ, Kellum JA, Plumb J, Mythen MG, Grocott MPW, Edwards MR, Miller TE; Perioperative Quality Initiative-3 workgroup; POQI chairs; Miller TE, Mythen MG, Grocott MP, Edwards MR; Physiology group; Preoperative blood pressure group; Intraoperative blood pressure group; Postoperative blood pressure group. Perioperative Quality Initiative consensus statement on intraoperative blood pressure, risk and outcomes for elective surgery. Br J Anaesth. 2019 May;122(5):563-574. doi: 10.1016/j.bja.2019.01.013. Epub 2019 Feb 27. PMID 30916004